CLINICAL TRIAL: NCT01638130
Title: Experiences and Needs of Patients With a High-grade Glioma and Their Caregivers
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: B322201110320
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Brain Neoplasms, Primary Malignant
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to explore the experiences and needs of patients with a high-grade glioma and their caregivers. Semi-structured interviews with patients and caregivers will be conducted and analysed using Grounded-Theory approach.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Patients with a primary high-grade glioma who are treated with chemo or were treated with chemo
* Caregivers of patients with a primary high-grade glioma who are treated with chemo or were treated with chemo
* Able to be interviewed
* Dutch

Exclusion Criteria:

* Patients with cerebral metastases
* Patients and caregivers who withdraw their informed consent
* Emotionally and cognitive not being able to be interviewed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a high-grade glioma and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-02 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium